CLINICAL TRIAL: NCT07329257
Title: Investigating Phenotypic, Epigenetic, and NeuroGenetic Traits in Rare and Ultra-rare Neurodevelopmental Disorders
Brief Title: Investigating Phenotypic, Epigenetic, and NeuroGenetic Traits in Rare and Ultra-rare Neurodevelopmental Disorders (Project PENGUIN)
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, William David Arnold, Executive Director, UM System NextGen Precision Health Initiative. Professor, Physical Medicine and Rehabilitation, University of Missouri-Columbia
Other Study IDs: 2130290; SYT-1 (Registry Identifier: Synaptotagmin 1-Associated Neurodevelopmental Disorder)
Record Dates: First submitted 2025-12-10; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Baker Gordon Syndrome; Rare Neurodevelopmental Conditions; Rare Neurogenetic Conditions; Syt-1 Disorder; Epilepsy; Seizure; Genetic Mutations; Autism in Children; Developmental Delay (Disorder)
Keywords: Baker Gordon Syndrome; BAGOS; Rare Conditions; Rare; Neurogenetic; Neurodevelopmental; Ultra-rare; Genetic mutation; Autism
MeSH Terms: conditions — Epilepsy; Seizures; Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants in this study have the option to provide a one-time skin biopsy and/or blood draw.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — There is no intervention for this Natural History Study

SUMMARY:
Rare genetic neurodevelopmental disorders, such as Syt-1 or Baker Gordon Syndrome (BAGOS) arise from mutations in genes essential for brain development and function, often disrupting neurotransmission and neuronal connectivity. These conditions present with a wide range of symptoms including developmental delays, seizures, motor and behavioral challenges, and vary widely in severity. These disorders are complex, and they remain poorly understood and lack effective treatments.

Natural history and clinical genetic studies are crucial for mapping how these disorders progress, improving diagnostic accuracy, and guiding therapy development. A major focus is identifying reliable biomarkers (genetic, imaging, and physiological) to track disease severity and support clinical trials. This study will securely collect and analyze data to better understand disease impact, develop patient-derived model systems, and build resources to support future treatments.

DETAILED DESCRIPTION:
Rare genetic neurodevelopmental disorders are a diverse group of conditions caused by mutations in genes critical to brain development and function. These disorders often involve disruptions in key proteins responsible for processes like neurotransmitter release, synaptic signaling, and neuronal connectivity. For example, mutations in genes such as SYT1 (which encodes synaptotagmin-1, a calcium-sensing protein essential for regulated neurotransmission) can lead to severe conditions like SYT1-associated neurodevelopmental disorder, also known as Baker-Gordon Syndrome (BAGOS). Similar mutations in other genes may result in distinct but overlapping clinical syndromes.

These rare disorders typically present with a wide range of symptoms, including developmental delays, intellectual disability, seizures, abnormal motor function, behavioral changes, visual impairments, and in some cases, self-injurious behaviors. The severity and progression of symptoms can vary significantly between individuals, even among those with the same genetic diagnosis.

Due to their rarity and complexity, many of these conditions are poorly understood, and treatment options remain limited. Therefore, natural history studies and clinical genetic studies play a crucial role in advancing research. These studies systematically collect data over time to understand how symptoms evolve, how quickly the disease progresses, and what measurable changes occur in affected individuals.

A key component of studies in rare genetic diseases is the identification and validation of biomarker quantifiable indicators such as genetic signatures, brain imaging findings, or physiological measurements-that can serve as reliable endpoints in clinical trials. By tracking these markers, researchers can better evaluate the efficacy of potential therapies and design more targeted treatments.

In addition to guiding drug development, these studies help researchers recognize broader patterns across neurodevelopmental disorders. This can lead to the discovery of undiagnosed cases, improve diagnostic accuracy, and foster earlier intervention. Ultimately, building a comprehensive understanding of these rare genetic conditions is essential for improving quality of life for affected individuals and their families. The investigators will analyze this information to explore how rare neurodevelopmental disorders affect ongoing neurodevelopment and quality of life. This study aims to lay groundwork for future therapies and will improve our understanding of rare neurogenetic disorders.

ELIGIBILITY:
For those with a rare condition:

Inclusion Criteria:

* Diagnosed or suspected neurogenetic disorder
* Individuals 0-99

Exclusion Criteria:

* Individuals unwilling or unable to complete visits with the study team.

For control parents/caregivers of those with a rare condition:

Inclusion Criteria:

* No history of a neurological disorder.
* >18 years.
* Legal caregiver of the patient diagnosed with a rare neurodevelopmental disorder.

Exclusion Criteria:

* Individuals unwilling or unable to complete the visit with the study team.
* Individuals who have a history of neurological disorders.
* < 18 years old

For all individuals who participate in the skin biopsy:

* Individuals with disease that is known to be associated with poor wound healing.
* Individuals with a history of allergic reaction to lidocaine.
* Medical History of cellulitis, diabetes mellitus, poor extremity circulation, deep vein thrombosis, or a history of non-traumatic amputation.
* Currently taking anticoagulation or have taken with last 6 months

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosed or suspected rare genetic neurodevelopmental disorder. Parents and caregivers over 18 years of age can participate in the study as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease onset patterns, symptom evolution, and progression severity in rare neurodevelopmental disorders | 3 years
Identify and validate biomarkers (genetic, imaging, and physiological) that correlate with disease severity and progression | 3 years
Establish patient-derived and control cell lines (e.g., fibroblasts, induced pluripotent stem cells) to generate model systems for mechanistic studies and pre-clinical evaluation of potential therapies | 3 years

SECONDARY OUTCOMES:
Develop a deep phenotypic profile (cognitive, motor, behavioral, and neurological) | 3 years
  Functional Mobility Scale, Aberrant Behavior Checklist, Conners Global Index, Pediatric Sleep Questionnaire, Medical Questionnaires, Ex.
Distribution of clinical presentation features, including age at onset, core symptoms, severity scores, and disease progression measures, within and across genetic subtypes | 3 years
Build a repository to support future interventional clinical trials | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: W. David Arnold, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No